CLINICAL TRIAL: NCT06675799
Title: Sleep Extension to Improve Mood in Young Urban Adults
Brief Title: Pilot Sleep Extension and Mood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1230
Record Dates: First submitted 2024-10-28; First posted 2024-11-05 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-02

CONDITIONS: Internalizing Mental Health Symptoms; Sleep Problems
Keywords: young adults; sleep; mood; anxiety; depression; sleep extension; stress
MeSH Terms: conditions — Parasomnias; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Extension (Experimental): Sleep-related psychoeducation will be provided in weekly lesson content. Phone coaching will revolve around sleep health and meeting sleep goals.
  Interventions: Behavioral: Sleep Extension
- Healthy Living (Active Comparator): Psychoeducation about general health (e.g., hand washing) will be provided in weekly lesson content. Phone coaches will not provide counseling or goal setting but may clarify terms or concepts.
  Interventions: Behavioral: Healthy Living Psychoeducation

INTERVENTIONS:
Behavioral: Sleep Extension — Weekly educational material about sleep health and weekly brief phone coaching calls for a total of 6 weeks.
  Arms: Sleep Extension
Behavioral: Healthy Living Psychoeducation — Weekly educational materials about healthy habits and weekly brief phone calls to clarify terms or concepts.
  Arms: Healthy Living

SUMMARY:
The goal of this interventional study is to learn if a digital sleep extension intervention can improve sleep and mood in young urban adults with mood symptoms. The main questions it aims to answer are:

Will this intervention improve sleep? Will this intervention improve mood? Does the effect of this intervention change based on environmental factors like noise and light pollution?

Researchers will compare participants receiving the sleep intervention to participants receiving a "general healthy living" intervention to see if outcome are different across groups.

Participants will:

* receive 6 weeks of brief once weekly telephone coaching and read once weekly educational content
* have their sleep monitored daily with a FitBit and Somnofy sleep device and during the 6-week intervention period
* respond to questionnaires at the start of the intervention, halfway through the intervention, at the end of the intervention, and finally 4 weeks after completing the intervention

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 30
* Have internalizing symptoms (e.g., depression, anxiety, stress)
* Have sleep concerns
* Sleep less than 7 hours per night
* Have perceived neighborhood disorder
* Smart phone that can run Somnofy app
* Access to Wifi in their home

Exclusion Criteria:

* High risk for obstructive sleep apnea
* Significant medical morbidities or psychiatric problem, or chronic substance use
* Non-English speaking (unable to participate in therapy or questionnaire)
* Taking medications for sleep
* An insomnia disorder
* Traveling for 2 weeks or more during the 10-week study period (due to loss of data from participants not sleeping in their home where the Somnofy device has been set up)
* Employed with rotating shift or night work

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Feasibility | From enrollment to the end of post-treatment follow-up period (10 weeks after start of intervention)
  Measured by the number of participants approached, recruited and retained
Tolerability | From enrollment to the end of post-treatment follow-up period (10 weeks after start of intervention)
  Measured by sessions completed
Acceptability | At end of 6-week intervention
  Acceptability of Intervention Measure
Sleep duration | From enrollment to the end of post-treatment follow-up period (10 weeks after start of intervention)
  Measured by Fitbit
Sleep efficiency | From enrollment to the end of post-treatment follow-up period (10 weeks after start of intervention)
  Measured by Fitbit
Waking after sleep onset (WASO) | From enrollment to the end of post-treatment follow-up period (10 weeks after start of intervention)
  Measured by Fitbit
Subjective sleep quality | From enrollment to the end of post-treatment follow-up period (10 weeks after start of intervention)
  Measured with the Pittsburgh Sleep Quality Index (PSQI), where higher scores indicate poorer sleep quality.
Internalizing symptoms | From enrollment to the end of post-treatment follow-up period (10 weeks after start of intervention)
  Anxiety, depression, and stress as measured with the Depression, Anxiety and Stress Scale - 21 item (DASS-21), where higher scores mean more distress.

SECONDARY OUTCOMES:
Daytime fatigue | From enrollment to the end of post-treatment follow-up period (10 weeks after start of intervention)
  PROMS-Fatigue 8 item
Bedtime Procrastination | From enrollment to the end of post-treatment follow-up period (10 weeks after start of intervention)
  Bedtime Procrastination Scale where higher scores equal more procrastination.
Electronics use before bed | Pre-treatment and at 6-week post-treatment assessment
  2 items taken from National Sleep Foundation 2011 Sleep in America survey

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Duffecy, PhD, Principal Investigator — University of Illinois Chicago
Locations (1):
- University of Illinois Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided